CLINICAL TRIAL: NCT06098144
Title: Expanding the Role of the Safety Manager to Implement a Workplace Smoking Cessation Program in the Construction Sector
Brief Title: Smoking Cessation Program in the Construction Sector
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Principal Investigator, Taghrid Asfar, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230549
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation; Tobacco Use Cessation; Tobacco Smoking
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Tobacco Smoking | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: Cluster-randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 Group A: Tobacco Quit-line (TQL) Group (Experimental): Participants will be referred to the TQL and will be followed up for up to 12 months.
  Interventions: Behavioral: Tobacco Quit-line
- Phase 1 Group B: Brief Behavioral Counseling Group (Experimental): Participants will receive one brief behavioral counseling session and two phone call follow-ups, then be followed up for 12 months. Besides the counseling session, they will be provided with Nicotine Replacement Therapy (NRT) and a referral to the TQL.
  For the NRT, participants will receive one box of Nicorette nicotine gums, 2 mg or 4 mg (depending on the number of cigarettes smoked), as well as 8 additional gums for a total of 168 gums during the counseling session. This amount is enough for 3 weeks. An additional 3-week supply will be provided at the second follow-up.
  Interventions: Drug: Nicorette; Behavioral: Tobacco Quit-line; Behavioral: Brief Behavioral Counseling
- Phase 2 Group A: Second Tobacco Quit-line (TQL) Group (Experimental): Participants from Group A who did not quit smoking at the 3-month follow-up may receive a second referral to the TQL and will be followed up for up to 12 months.
  Interventions: Behavioral: Tobacco Quit-line
- Phase 2 Group B: Second Brief Behavioral Counseling Group (Experimental): Participants from Group B who did not quit smoking at the 3-month follow-up may receive a second brief behavioral counseling session and two phone call follow-ups, then be followed up for 12 months. Besides the counseling session, they will be provided with Nicotine Replacement Therapy (NRT) and a second referral to the TQL.
  For the NRT, participants will receive one box of Nicorette nicotine gums, 2 mg or 4 mg (depending on the number of cigarettes smoked), as well as 8 additional gums for a total of 168 gums during the counseling session. This amount is enough for 3 weeks. An additional 3-week supply is provided at the second follow-up.
  Interventions: Drug: Nicorette; Behavioral: Tobacco Quit-line; Behavioral: Brief Behavioral Counseling
- Phase 2 Group A + C: TQL and Intensive Behavioral Counseling Group (Experimental): Participants from Phase 1 Group A who did not quit smoking at the 3-month follow-up may receive four behavioral counseling sessions, two phone-call follow-ups, and Nicotine Replacement Therapy (NRT) and be followed up for 12 months.
  For the NRT, participants will receive one box of Nicorette nicotine gums, 2 mg or 4 mg (depending on the number of cigarettes smoked), as well as 8 additional gums for a total of 168 gums during the first counseling session. This amount is enough for 3 weeks. An additional 3-week supply is provided at the fourth session.
  Interventions: Drug: Nicorette; Behavioral: Tobacco Quit-line; Behavioral: Intensive Behavioral Counseling
- Phase 2 Group B + C: Brief Counseling and Intensive Behavioral Counseling Group (Experimental): Participants from Phase 1 Group B who did not quit smoking at the 3-month follow-up may receive four behavioral counseling sessions, two phone-call follow-ups, and Nicotine Replacement Therapy (NRT) and be followed up for 12 months.
  For the NRT, participants will receive one box of Nicorette nicotine gums, 2 mg or 4 mg (depending on the number of cigarettes smoked), as well as 8 additional gums for a total of 168 gums during the first counseling session. This amount is enough for 3 weeks. An additional 3-week supply is provided at the fourth session.
  Interventions: Drug: Nicorette; Behavioral: Tobacco Quit-line; Behavioral: Brief Behavioral Counseling; Behavioral: Intensive Behavioral Counseling

INTERVENTIONS:
Drug: Nicorette — Participants will receive a 6-week supply of nicotine replacement treatment (NRT). Based on participants' self-report on the number of cigarettes smoked, these are the possible dosages of NRT gum (2 mg and 4 mg). Participants should not smoke and use the nicotine gum at the same time. Nicotine gum should only be used when cravings for cigarettes arise and should not be treated like regular chewing gum. It is not to be constantly chewed
  NRT will be distributed based on the treatment condition.
  Arms: Phase 1 Group B: Brief Behavioral Counseling Group; Phase 2 Group A + C: TQL and Intensive Behavioral Counseling Group; Phase 2 Group B + C: Brief Counseling and Intensive Behavioral Counseling Group; Phase 2 Group B: Second Brief Behavioral Counseling Group
Behavioral: Tobacco Quit-line — The TQL is free, and the TQL counselor will provide three phone counseling sessions lasting approximately 15 minutes to devise a specific plan to quit smoking and arrange the delivery of 4 to 12 weeks of NRT based on need. Participants will be advised to request nicotine gums instead of patches to accommodate their job circumstances.
Behavioral: Brief Behavioral Counseling — The counseling session will discuss preparing to quit, coping with job-related stress, getting social support, the "5A's" for preventing relapse (Avoid, Alter, Alternatives, Anticipate, and Active), proper use of NRT, and last approximately 30 minutes.
  Arms: Phase 1 Group B: Brief Behavioral Counseling Group; Phase 2 Group B + C: Brief Counseling and Intensive Behavioral Counseling Group; Phase 2 Group B: Second Brief Behavioral Counseling Group
Behavioral: Intensive Behavioral Counseling — Participants will receive four weekly counseling sessions which include information about how to quit, challenges, and short and long-term relapse prevention. Each session will last approximately 20 minutes.
  Arms: Phase 2 Group A + C: TQL and Intensive Behavioral Counseling Group; Phase 2 Group B + C: Brief Counseling and Intensive Behavioral Counseling Group

SUMMARY:
The main objective of this study is to identify the optimal adaptive smoking cessation program for the construction sector in terms of effectiveness, cost-effectiveness, and potential implementation.

ELIGIBILITY:
Inclusion Criteria:

Company leaders:

* ≥ 18 years
* Involved in decision making
* Willing to participate in the implementation development and evaluation

Safety Managers:

- ≥ 18 years Self-identified as a safety manager or superintendent Have no plans to leave the company in the next year Speak either English or Spanish Non-cigarette smoker Willing to receive training in smoking cessation treatment Willing to deliver the smoking cessation treatment to workers

Construction Workers:

* Be a construction worker
* ≥ 18 years
* Have smoked on average 5 or more cigarettes daily for the past year
* Willing to make a serious quit attempt in the next 30 days
* Willing to receive treatment from the Florida Tobacco Quitline.
* Planning to stay in the company for the next 6 months
* Own a telephone and plan to keep it active for the next 12 months

Exclusion Criteria:

Safety Managers:

- Current cigarette smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Program Effectiveness Measure in Percentage | Up to 4 years
  Will be collected as the difference in percentage of participants who quit smoking at the 12-month follow-up assessment between the three treatment groups.
Program Cost-Effectiveness Measured by Number of U.S Dollars | Up to 4 years
  Will be measured as the difference in the number of U.S. dollars between the three programs.
Program Cost-Effectiveness Measured by Quality Adjusted Life Years | Up to 4 years
  Will be measured by quality-adjusted life years defined as the difference in the number of years lived in perfect health between the three programs.

SECONDARY OUTCOMES:
Program's Implementation- Acceptability Measured by Likert Scale | Up to 4 years
  Using the Acceptability of Intervention Measure, acceptability will be scored on a 5-point Likert scale, with higher scores indicating greater acceptability.
Program's Implementation- Feasibility Measured by Likert Scale | Up to 4 years
  Using the Feasibility of Intervention Measure, feasibility will be scored on a 5-point Likert scale, with higher scores indicating greater feasibility.
Program's Implementation- Sustainability Measured by Likert Scale | Up to 4 years
  Using the Intervention Sustainability Assessment Tool, sustainability will be scored on a 7-point Likert scale, with higher scores indicating greater sustainability.

CONTACTS AND LOCATIONS:
Overall Officials: Taghrid Asfar, MD, Principal Investigator — tasfar@miami.edu
Locations (1):
- Don Soffer Clinical Research Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asfar T, Lee DJ, Salloum RG, LeLaurin JH, Kobetz E, Pradhananga N, De Dios Despaux RA, McCollister KE, Oluwole O, Corbin L, Laine J, Bursac Z. Empowering safety managers to champion the implementation of smoking cessation services in the construction industry: Protocol for a sequential multiple assignment randomized trial. PLoS One. 2025 Jun 9;20(6):e0324717. doi: 10.1371/journal.pone.0324717. eCollection 2025. PMID 40489501

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT06098144/Prot_SAP_001.pdf